CLINICAL TRIAL: NCT05504707
Title: Phase 1 Dose-Escalation, Dose-Expansion Trial of Intratumoral HER2- and HER3-Primed Dendritic Cells Injections for the Treatment of Early-Stage TNBC and ER Low Positive Breast Cancer (DecipHER)
Brief Title: DecipHER Trial - DC1 Tx for Early-Stage TNBC and ER Low Positive Breast Cancer
Acronym: DecipHER
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: H. Lee Moffitt Cancer Center and Research Institute (Other)
Collaborators: The Shulas' Foundation (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: MCC-20897
Record Dates: First submitted 2022-08-15; First posted 2022-08-17 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-02

CONDITIONS: Triple Negative Breast Cancer; HER2-negative Breast Cancer
Keywords: Breast Cancer
MeSH Terms: conditions — Triple Negative Breast Neoplasms; Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Dendritic Cell Vaccine dose Escalation (Experimental): Dose escalation to determine the maximum tolerated dose (MTD) of HER2- and HER3- primed DC1 study vaccines. Participants will be treated in cohorts of size three to six and the dosage will be escalated if the clinical toxicity is acceptable. A total of 3 dose levels will be used.
  Interventions: Biological: HER2 - primed Dendritic cells; Biological: HER3 - primed Dendritic cells

INTERVENTIONS:
Biological: HER2 - primed Dendritic cells — Dendritic cell will be administered at ultra-sound guided injections. Participants will receive 8 intratumoral injections. These injections will be administered twice per week per week (given 3 days apart). Participants will receive alternating injections (3 days apart) of HER2-primed followed by HER3-primed DCs.
  Participants will be treated at the following dose levels:
  Dose level 1: HER2 - primed Dendritic cells dose 10-20 million Dose level 2: HER2 - primed Dendritic cells dose 30-50 million Dose level 3: HER2 - primed Dendritic cells dose 80-100 million
Biological: HER3 - primed Dendritic cells — Dendritic cell will be administered at ultra-sound guided injections. Participants will receive 8 intratumoral injections. These injections will be administered twice per week per week (given 3 days apart). Participants will receive alternating injections (3 days apart) of HER2-primed followed by HER3-primed DCs.
  Participants will be treated at the following dose levels:
  Dose level 1: HER3 - primed Dendritic cells dose 10-20 million Dose level 2: HER3 - primed Dendritic cells dose 30-50 million Dose level 3: HER3 - primed Dendritic cells dose 80-100 million

SUMMARY:
The purpose of the study is to find out if an investigational vaccine called Dendritic Cell (DC) vaccine given together with standard of care chemotherapy drugs can help people with Triple Negative and HR low positive breast cancer.

ELIGIBILITY:
Inclusion Criteria:

* A diagnosis of HER2-negative breast cancer.
* Diagnosis of HR negative or HR low positive tumor.
* Clinical stage T1c, nodal stage N1-N2 or stage T2-4, nodal stage N0-N2 breast cancer.
* Participant must be medically and surgically appropriate to undergo neoadjuvant chemotherapy regimen followed by standard of care local therapy as determined by their treating physician.
* Age ≥18 years.
* ECOG performance status 0 or 1.
* Patients must have normal organ and marrow function, as defined below, within 14 days of registration:
* *Absolute neutrophil count (ANC) ≥ 1500/μL
* *Platelets ≥ 75 000/μL
* *Total bilirubin ≤ 1.5 x institutional ULN, except patients with Gilbert's syndrome in whom total bilirubin must be < 3.0 mg/dL
* *AST/ALT ≤ 3 x institutional ULN
* *Creatinine ≤ 1.5 x institutional ULN
* Left ventricular ejection fraction above institutional lower limit of normal (by echocardiogram or MUGA scan).
* Female patients of childbearing potential must agree to use dual methods of contraception and have a negative serum pregnancy test at screening. Acceptable methods of contraception are condoms with contraceptive foam, oral, implantable or injectable contraceptives, contraceptive patch, intrauterine device, diaphragm with spermicidal gel, or a sexual partner who is surgically sterilized or post-menopausal. Effective methods of contraception must be used throughout the study and for 5 months following the last dose. To show that women do not have childbearing potential, postmenopausal women must be amenorrheic for at least 12 months naturally (and not because of/following chemotherapy) or patients must be surgically sterile.
* Ability to understand and the willingness to sign a written informed consent agreement prior to study registration.

Exclusion Criteria:

* Patients who received prior anthracycline-based chemotherapy for the treatment of any cancer.
* Patients with inflammatory breast cancer.
* Patients must not be receiving any other investigational agents or active antineoplastic therapies.
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
* Patients with active autoimmune disease or history of autoimmune disease that might recur, which may affect vital organ function or require immune-suppressive treatment, including chronic prolonged systemic corticosteroid use (defined as corticosteroid use lasting one month or more).
* Female patients who are pregnant or nursing.
* No other prior malignancy is allowed, except for the following: a. adequately treated basal-cell or squamous-cell skin cancer, b. in situ cervical cancer, c. or any other cancer from which the patient has been disease free for at least 3 years.
* History of testing positive for human immunodeficiency virus (HIV) or acquired immunodeficiency syndrome (AIDS).
* History of positive test for Hepatitis B or Hepatitis C virus indicating acute or chronic infection.
* Patients who have received a live attenuated vaccine ≤ 30 days prior to registration.
* Unable to comply with the treatment schedule and study procedures for any reason.
* Previously treated with breast cancer-directed vaccine therapies in prior 3 months.
* Previously treated with any form HER2- or HER3-primed DC1 therapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2022-08-26 (Actual); Primary Completion 2026-10 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
Maximum Tolerated Dose (MTD) | 4 weeks after start of treatment
  Maximum Tolerated Dose (MTD) of HER2- and HER3- primed DC1 study vaccines. The MTD will be defined as the highest dose level at which < 2 of 6 patients experience dose-limiting toxicities (DLTs).

SECONDARY OUTCOMES:
Number of Dose Limiting Toxicities | 5 weeks after start of treatment
  Number of DLTs experienced by participants
Participants with pathological complete response after receiving HER2/HER3 DC1 intratumoral injections | Up to 24 weeks
  Pathological complete response defined as the absence of invasive breast cancer in the breast and lymph nodes after completion of treatment with DC1 injections and neoadjuvant chemotherapy.
Participants with clinical and radiological responses after receiving HER2/HER3 DC1 | Up to 36 Months
  Clinical or radiological complete responses (CR): Palpable or visible lesion(s) identified at baseline are no longer palpable and there are no new lesion(s) or other signs of disease progression.
Participants with clinical and radiological partial responses after receiving HER2/HER3 DC1 | Up to 36 Months
  Clinical or radiological partial responses (PR): A reduction in the product of the two largest perpendicular diameters of the primary tumor by 50% or more.
Participants with clinical and radiological progression of disease after receiving HER2/HER3 DC1 | Up to 36 Months
  Clinical or radiological progression of disease (PD): An increase in the product of the two largest perpendicular diameters of the primary tumor by 25% or more or the presence of a new lesion.
Participants with clinical and radiological stable disease after receiving HER2/HER3 DC1 | Up to 36 Months
  Clinical or radiological stable disease (SD): Neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD.
Participants with Recurrence Free Survival (RFS) | Up to 36 Months
  Recurrence free survival (RFS) defined as time I months to breast cancer recurrence or death (whichever comes first) since date of surgical treatment of breast cancer.

CONTACTS AND LOCATIONS:
Overall Officials: Ricardo Costa, MD, Principal Investigator — Moffitt Cancer Center
Locations (1):
- Moffitt Cancer Center, Tampa, Florida, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: Moffitt Clinical Trial Search — https://moffitt.org/clinical-trials-research/clinical-trials/?gclid=EAIaIQobChMImIymzIa-9gIVAZ2GCh3uzAWJEAAYASAAEgI0ovD_BwE